CLINICAL TRIAL: NCT04267211
Title: Prenatal Consult With Illustrated Literature
Acronym: PNCIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Swanson, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19892
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Premature Birth; Prenatal Stress
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Illustrated Consult (Experimental)
  Interventions: Other: Illustrated handout at prenatal consult
- Standard Consult (Experimental)
  Interventions: Other: Standard Prenatal Consult

INTERVENTIONS:
Other: Illustrated handout at prenatal consult — Illustrated consult group will be given an illustration paper describing the majority of the issues discussed at the prenatal consult
  Arms: Illustrated Consult
Other: Standard Prenatal Consult — Standard prenatal consult
  Arms: Standard Consult

SUMMARY:
The overall purpose of this study is to determine whether implementing a 'Prenatal Consult Bundle' to the existing prenatal consult, including provision of sample questions, added discussion points and handouts, and a return visit, will decrease parental anxiety and improve information recall. Additionally, this study will determine if this effect is further increased with the use of illustrated literature.

DETAILED DESCRIPTION:
This study will be a prospective randomized control trial. Seventy participants will be enrolled for the 'Standard' consult. These women will receive a questionnaire 6-24 hours after their consult. Then 140 participants will be randomized to either the 'Standard Upgrade' or 'Illustrated Upgrade' arm. Randomization will additionally be stratified based on estimated gestational age. These participants will receive an upgraded consult implementing the 'Prenatal Consult Bundle' which emphasizes the parents' role and follow up, with or without an illustrated handout. These participants will receive the same questionnaire 6-24 hours after their consult. Demographic information collected will include maternal age, gravidity, use of magnesium, social support and health literacy. All data will be collected to assess whether either arm of the consult 'upgrade' reduces anxiety or improves knowledge retention after the prenatal consult. Analyses will be completed using Statistical Analysis Software (SAS) using appropriate statistical testing.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women admitted to OB unit at the University of Virginia Medical Center
* Estimated gestational age of >25 weeks and <35 weeks

Exclusion Criteria:

* Non-English Speaking
* Pregnant women <15 years of age
* Known critical conditions or congenital anomalies
* Women who have had any prior prenatal consultations regarding current pregnancy

Ages: 15 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Maternal Anxiety | Within 48 hours of consultation
  Using the State-Trait Anxiety Inventory (STAI), maternal anxiety will be assessed between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Namrita Odackal, MD, Principal Investigator — University of Virginia
Locations (1):
- UVA Health, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Odackal NJ, Conaway M, Cha J, Swanson JR. Prenatal consults with illustrated literature (PnCIL): a RCT studying visual aids during prenatal consults. J Perinatol. 2020 Aug;40(8):1154-1162. doi: 10.1038/s41372-020-0709-y. Epub 2020 Jun 8. PMID 32514007